CLINICAL TRIAL: NCT05325346
Title: A Phase I, Open-Label, Randomized, Three-Period, Three-Sequence Crossover Study of the Effects of Co-administration of Intravenous VLX-1005 With Argatroban on Pharmacokinetics, Pharmacodynamics and Safety in Healthy Adult Subjects
Brief Title: A Phase I Study of the Co-administration of VLX-1005 and Argatroban in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Veralox Therapeutics (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VLX-1005-002
Record Dates: First submitted 2022-03-04; First posted 2022-04-13 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-03

CONDITIONS: Heparin-induced Thrombocytopenia
MeSH Terms: interventions — argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VLX-1005 (Experimental): Intravenous administration of VLX-1005 with measurements of PK and PD
  Interventions: Drug: VLX-1005
- Argatroban (Active Comparator): Intravenous administration of argatroban with measurements of PK and PD
  Interventions: Drug: Argatroban
- VLX-1005 and Argatroban (Other): Intravenous co-administration of VLX-1005 and argatroban with measurements of PK and PD
  Interventions: Drug: VLX-1005; Drug: Argatroban

INTERVENTIONS:
Drug: VLX-1005 — Measurement and comparison of the effects and potential interactions between VLX-1005 and argatroban on safety, tolerability, PK and PD
  Arms: VLX-1005; VLX-1005 and Argatroban
Drug: Argatroban — Measurement and comparison of the effects and potential interactions between VLX-1005 and argatroban on safety, tolerability, PK and PD
  Arms: Argatroban; VLX-1005 and Argatroban

SUMMARY:
The study is designed to characterize the safety and tolerability of VLX-1005 and argatroban administered intravenously, either alone or in combination; and the pharmacokinetics and pharmacodynamics and potential interaction of both agents in a population of healthy subjects.

DETAILED DESCRIPTION:
VLX-1005 is being developed as a treatment for heparin induced thrombocytopenia (HIT), a rare but life threatening illness. Currently, the anticoagulant argatroban remains the standard of care for treating HIT. However, this treatment remains inadequate due to both thrombosis and major bleeding complications that each may exceed 30% of treated HIT patients. These findings are significant to the later stage clinical development of VLX-1005 as a trial of VLX-1005 on top of argatroban therapy would require an understanding of any potential drug-drug interactions- whether direct or via metabolism. Specifically, coadministration of VLX-1005 with argatroban mandates an analysis of the potential effects on PK, pharmacodynamics and bleeding. The current study is designed to address these important questions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (non-lactating and not of childbearing potential) subjects age 19 to 55 inclusive.
2. Females must have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

   1. hysteroscopic sterilization
   2. bilateral tubal ligation or bilateral salpingectomy
   3. hysterectomy
   4. bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
3. Good general health, with no significant medical history. Subjects must have no clinically significant abnormalities at screening, and/or before administration of the initial dose of study drug.
4. Body weight ≥ 50 kg at the screening visit.
5. Body Mass Index (BMI) between 18 and 32 kg/m2 inclusive.
6. Laboratory values (clinical chemistry and hematology) within the normal reference range. Deviations from this range may be acceptable if they are considered 'not clinically significant' (NCS) by the PI, however, AST and ALT shall be <1.5x ULN. 7. Males who have not been vasectomized prior to participating in the study must agree to use at least 2 approved methods of contraception, or to abstain from sexual intercourse, from randomization until 90 days after their last dose of VLX-1005 and should refrain from donating sperm during that period. 8. Is a non-smoker and must not have used any nicotine products within three months prior to screening.

9. Able and willing to attend the necessary visits to the study center.

Exclusion Criteria:

1. Blood donation or recipient of blood transfusion in previous 12 weeks.
2. History of clinically significant endocrine, neurological, gastrointestinal, cardiovascular, hematological, hepatobiliary, immunological, renal, respiratory, or genitourinary abnormalities or diseases.
3. History of neoplastic disease (with the exception of adequately treated nonmelanomatous skin carcinoma).
4. Mentally or legally incapacitated (e.g. has significant emotional problems at the time of Screening Visit or expected during the conduct of the study, or has a history of a clinically significant psychiatric disorder within the last 5 years).
5. Fever (body temperature >38 C) or symptomatic viral/bacterial infection or use of antibiotics within 2 weeks prior to Screening.
6. Supine resting blood pressure (BP) >140/90 mmHg or heart rate (HR) >100 beats per minute at Screening and at Day -2.
7. Clinically significant abnormality on ECG performed at the Screening Visit or prior to administration of the initial dose of study drug. (Abnormalities include not being in sinus rhythm, IVCD/BBB or QTcF>450 ms for males (470 ms for females)).
8. Out of range (on repeat) testing for coagulation tests.
9. Clinically significant laboratory abnormalities including: Impaired renal function (estimated creatinine clearance (CrCl) of <80 mL/minute based on CrCl = (140-age [years])(body weight [kg])/(72)(serum creatinine [mg/dL])).
10. Positive test for hepatitis C antibody, hepatitis B surface antigen, or human immunodeficiency virus (HIV) antibody at Screening.
11. Participants with a positive toxicology screening panel (urine test including qualitative identification of barbiturates, tetrahydrocannabinol, amphetamines, benzodiazepines, opiates, cocaine, cotinine and ethanol).
12. Participants with a history of substance abuse or dependency or history of recreational IV drug use (by self-declaration).13. Participant has a suspected history of alcohol abuse in the 6 months prior to screening.

14. Use of NSAIDs, aspirin or aspirin-containing medications (and other medications affecting platelet function [for example cilostazol, clopidogrel, ticagrelor, prasugrel, dipyridamole]) in the 14 days prior to dosing with study medication. VerifyNow testing will be performed at check-in to exclude possible use of medications that affect platelet function.

15. Unable to refrain from or anticipates the use of any medications, including prescription and non-prescription drugs and herbal remedies (such as St. John's Wort [Hypericum perforatum]), beginning 14 days (or 5 half-lives, whichever is longer) before administration of the initial dose of study drug and continuing throughout the study until the final study visit. There may be certain medications that are permitted at the discretion of the PI and Sponsor (including paracetamol/acetaminophen, medications for the treatment of AEs following administration of study drug).

16. Subjects who are unlikely to comply with the study protocol or, in the opinion of the PI, would not be a suitable candidate for participation in the study.

17. Have participated in any other investigational drug trial within 30 days of dosing in the present study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Effects of argatroban on Cmax of VLX-1005 | 0 - 51 hours
  Measure the effects of argatroban on the maximum plasma concentration (Cmax) of VLX-1005
Effects of VLX-1005 on Cmax of argatroban | 0 - 51 hours
  Measure the effects of VLX-1005 on the maximum plasma concentration (Cmax) of argatroban
Effects of argatroban on Tmax of VLX-1005 | 0 - 51 hours
  Measure the effects of argatroban on the time to maximum plasma concentration (Tmax) of VLX-1005
Effects of VLX-1005 on Tmax of argatroban | 0 - 51 hours
  Measure the effects of VLX-1005 on the time to maximum plasma concentration (Tmax) of argatroban
Effects of argatroban on AUC(inf) of VLX-1005 | 0 - 51 hours
  Measure the effects of argatroban on the Area Under the Curve [AUC(inf)] of VLX-1005
Effects of VLX-1005 on AUC(inf) of argatroban | 0 - 51 hours
  Measure the effects of VLX-1005 on the Area Under the Curve [AUC(inf)] of argatroban
Effects of VLX-1005 on whole blood aggregometry | 0 - 9 hours
  The change in impedance from baseline by whole blood aggregometry will be measured to assess the effects of VLX-1005 on platelet aggregation
Effects of argatroban on whole blood aggregometry | 0 - 9 hours
  The change in impedance from baseline by whole blood aggregometry will be measured to assess the effects of argatroban on platelet aggregation
Effects of VLX-1005 on PFA-100 | 0 - 9 hours
  Change in PFA-100 (a platelet pharmacodynamic measure) from baseline, to assess the effects of VLX-1005 on platelet aggregation
Effects of argatroban on PFA-100 | 0 - 9 hours
  Change in PFA-100 (a platelet pharmacodynamic measure) from baseline, to assess the effects of argatroban on platelet aggregation

SECONDARY OUTCOMES:
Safety as measured by incidence of Treatment Emergent Adverse Events | 0 - 30 days
  To assess the effects on subject safety of VLX-1005 and argatroban alone and in combination as measured by incidence of Treatment Emergent Adverse Events as assessed by CTCAE, ver 5.0.
Effects of VLX-1005 on 12-HETE | 0 - 12 hours
  12-hydroxyeicosatetraenoic acid (12-HETE), a platelet biomarker, will be measured to assess the effects of VLX-1005 on its production
Effects of argatroban on 12-HETE | 0 - 12 hours
  12-HETE, a platelet biomarker, will be measured to assess the effects of argatroban on its production

CONTACTS AND LOCATIONS:
Overall Officials: Allen Hunt, MBA, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No